CLINICAL TRIAL: NCT00515619
Title: An International Open-label Extension Trial to Determine Safety and Efficacy of Long-term Oral Lacosamide (SPM 927) in Patients With Partial Seizures
Brief Title: Assess Safety and Efficacy of Lacosamide in Patients With Partial Seizures
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SP0774; 2004-000152-16 (EudraCT Number)
Record Dates: First submitted 2007-08-13; First posted 2007-08-14 (Estimated); Results first posted 2011-09-09 (Estimated); Last update posted 2017-08-28 (Actual); Status verified 2017-07

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — Lacosamide; 2-(acetylamino)-3-methoxy-N-(phenylmethyl)-, (2R)-

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lacosamide (Experimental): 50 mg and 100 mg tablets up to 800 mg/day as twice day (BID) dosing
  Interventions: Drug: Lacosamide

INTERVENTIONS:
Drug: Lacosamide — 50 mg and 100 mg tablets up to 800 mg/day as twice day (BID) dosing throughout the trial
  Other Names: SPM 927; LCM

SUMMARY:
The main purpose of this trial is to determine safety and efficacy of Lacosamide under long term therapy.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of Epilepsy
* completion of double blind trial

Exclusion Criteria:

* taking other investigational drug than Lacosamide
* meeting withdrawal criteria from double blind trial

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 376 (Actual)
Dates: Start 2004-12; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493
Locations (54):
- Australia (7):
  - Randwick, New South Wales
  - Maroochydore, Queensland
  - Woodville, South Australia
  - Clayton, Victoria
  - Parkville, Victoria
  - West Heidelberg, Victoria
  - Adelaide
- Zagreb, Croatia
- Czechia (6):
  - Brno
  - Hradec Králové
  - Olomouc
  - Ostrava-Trebovice
  - Pilsen
  - Prague
- Finland (4):
  - Helsinki
  - Kuopio
  - Oulu
  - Tampere
- France (5):
  - Lille
  - Lyon
  - Montpellier
  - Paris
  - Toulouse
- Germany (6):
  - Berlin
  - Erlangen
  - Göttingen
  - Marburg
  - München
  - Ulm
- Hungary (4):
  - Budapest
  - Pécs
  - Szeged
  - Szombathely
- Lithuania (2):
  - Kaunas
  - Vilnius
- Poland (4):
  - Bialystok
  - Gdansk
  - Krakow
  - Warsaw
- Russia (2):
  - Moscow
  - Saint Petersburg
- Spain (4):
  - Girona
  - Granada
  - Madrid
  - Zaragoza
- Sweden (3):
  - Gothenburg
  - Linköping
  - Stockholm
- United Kingdom (6):
  - Cardiff
  - Dundee
  - Glasgow
  - London
  - Salford
  - Swansea

REFERENCES:
- [Result] Borghs S, de la Loge C, Brabant Y, Cramer J. Sensitivity testing of the Seizure Severity Questionnaire (SSQ). Epilepsy Behav. 2014 Feb;31:281-5. doi: 10.1016/j.yebeh.2013.10.010. Epub 2013 Nov 22. PMID 24275520
- [Derived] Rosenow F, Kelemen A, Ben-Menachem E, McShea C, Isojarvi J, Doty P; SP774 study investigators. Long-term adjunctive lacosamide treatment in patients with partial-onset seizures. Acta Neurol Scand. 2016 Feb;133(2):136-144. doi: 10.1111/ane.12451. Epub 2015 Jul 2. PMID 26133811
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was started in December of 2004 with recruitment occurring in Australia, Croatia, Czech Republic, Finland, France, Germany, Hungary, Lithuania, Poland, Russia, Spain, Sweden, and the United Kingdom. The study had last patient last visit in August of 2010.
Pre-assignment Details: Safety Set consists of all subjects who received at least 1 dose of Lacosamide.
Groups:
- Lacosamide: 50 mg and 100 mg tablets of lacosamide up to 800 mg/day as twice day (BID) dosing throughout the trial (flexible dosing)
Period: Overall Study
Arm/Group | Lacosamide
Started | 376
Safety Set | 376
Completed | 160
Not Completed | 216
Not completed — Adverse Event | 34
Not completed — Lack of Efficacy | 92
Not completed — Withdrawal by Subject | 66
Not completed — Protocol Violation | 3
Not completed — Lost to Follow-up | 4
Not completed — Unsatisfactory compliance | 6
Not completed — Other: Site discontinuing trials | 2
Not completed — Other: Subject cannot attend visits | 2
Not completed — Other: Subject required surgery | 1
Not completed — Other: Subject moved to another country | 1
Not completed — Other: Investigator decision | 1
Not completed — Other: Subject became pregnant | 1
Not completed — Other: Request from sponsor | 1
Not completed — Other: Drug available on license | 1
Not completed — Other: Subject interested in other AED | 1

BASELINE CHARACTERISTICS:
Arm/Group | Lacosamide
Number analyzed (Participants) | 376
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 7
  Between 18 and 65 years | 366
  >=65 years | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.8 (11.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 169
  Male | 207
Region of Enrollment [Number; unit: participants]
  Finland | 16
  Spain | 26
  Lithuania | 42
  Russian Federation | 31
  United Kingdom | 20
  France | 10
  Czech Republic | 50
  Hungary | 31
  Poland | 37
  Croatia | 31
  Australia | 31
  Germany | 35
  Sweden | 16

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Reporting at Least 1 Treatment-emergent Adverse Event (TEAE) During the Treatment Period (up to 5.5 Years)
Description: Adverse events are any untoward medical occurrences in a subject administered study treatment, whether or not these events are related to treatment.
Time Frame: During the Treatment Period (up to 5.5 years)
Population: Of the 376 subjects who entered the study, 376 are included in this summary based on the Safety Set (SS). SS population: number of subjects treated.
Measure: Number; unit: Subjects
Arm/Group | Lacosamide
Number analyzed (Participants) | 376
Subjects | 311

2. Primary Outcome: Number of Subjects Prematurely Discontinuing Due to a Treatment-emergent Adverse Event (TEAE) During the Treatment Period (up to 5.5 Years)
Description: as for outcome 1
Time Frame: During the Treatment Period (up to 5.5 years)
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Lacosamide
Number analyzed (Participants) | 376
Subjects | 33

3. Primary Outcome: Number of Subjects Reporting at Least 1 Serious Adverse Event (SAE) During the Treatment Period (up to 5.5 Years)
Description: A serious adverse event is any untoward medical occurrences in a subject administered study treatment, whether or not the event is related to treatment, with at least one of the follow outcomes: death, life-threatening, initial inpatient hospitalization or prolongation of hospitalization, significant or persistent disability/incapacity, congenital anomaly/birth defect, or an important medical event that may jeopardize the subject and require a medical/surgical intervention.
Time Frame: During the Treatment Period (up to 5.5 years)
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Lacosamide
Number analyzed (Participants) | 376
Subjects | 87

4. Secondary Outcome: Median Percentage Change From Baseline in 28-day Seizure Frequency During the Treatment Period (up to 5.5 Years)
Description: Median percentage change is the median value with respect to the percent change from Baseline across the population of subjects. Percentage change is calculated as 100 times the difference of the seizure frequency for the treatment period and the Baseline seizure frequency divided by the baseline seizure frequency.
  Negative changes from Baseline indicate an improvement (i.e., a reduction) in 28-day seizure frequency.
Time Frame: Baseline, Treatment Period (up to 5.5 years)
Population: Of the 376 subjects who were enrolled/treated in the study, 376 are included in this summary based on the Full Analysis Set (FAS). FAS population: number of subjects treated with at least 1 post-baseline seizure diary day with available data during the SP774 study.
Measure: Median (Full Range); unit: Percentage change
Arm/Group | Lacosamide
Number analyzed (Participants) | 376
Percentage change | -49.9 [-100.0 to 422.8]

5. Secondary Outcome: Percentage of at Least 50% Responders During the Treatment Period (up to 5.5 Years)
Description: At least 50 percent response is based on the percentage reduction in 28-day seizure frequency during the Treatment Period of the open-label extension relative to the Baseline Phase of the prior study. This endpoint reflects the percentage of subjects with at least 50% reduction (ie, at least 50% change) in 28-day partial onset seizure frequency
Time Frame: Treatment Period (up to 5.5 years)
Population: as for outcome 4
Measure: Number; unit: Percentage of subjects
Arm/Group | Lacosamide
Number analyzed (Participants) | 376
Percentage of subjects | 50.0

ADVERSE EVENTS:
Time Frame: The adverse event summaries are based on data collected during the 5.5 years of the study for all 376 patients
Arm/Group | Lacosamide
Serious Adverse Events (participants affected / at risk) | 87/376
Other Adverse Events (participants affected / at risk) | 232/376
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lacosamide (N=376)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Exomphalos (Congenital, familial and genetic disorders) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 1 (1)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 (1)
Diplopia (Eye disorders) | 1 (1)
Scotoma (Eye disorders) | 1 (1)
Eye haemorrhage (Eye disorders) | 1 (1)
Anal fistula (Gastrointestinal disorders) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 1 (1)
Mechanical ileus (Gastrointestinal disorders) | 1 (1)
Chest pain (General disorders) | 2 (2)
Chest discomfort (General disorders) | 1 (1)
Hepatomegaly (Hepatobiliary disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Abscess limb (Infections and infestations) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1)
Postoperative wound infection (Infections and infestations) | 1 (1)
Intervertebral discitis (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Pilonidal cyst (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 3 (3)
Subdural haematoma (Injury, poisoning and procedural complications) | 3 (3)
Brain contusion (Injury, poisoning and procedural complications) | 3 (3)
Lower limb fracture (Injury, poisoning and procedural complications) | 3 (3)
Skin laceration (Injury, poisoning and procedural complications) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 1 (3)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Skull fracture (Injury, poisoning and procedural complications) | 1 (1)
Jaw fracture (Injury, poisoning and procedural complications) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1)
Skeletal injury (Injury, poisoning and procedural complications) | 1 (1)
Soft tissue injury (Injury, poisoning and procedural complications) | 1 (1)
Tooth fracture (Injury, poisoning and procedural complications) | 1 (1)
Weight decreased (Investigations) | 1 (1)
Electrocardiogram QT corrected interval prolonged (Investigations) | 1 (1)
Investigation (Investigations) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Brain neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Convulsion (Nervous system disorders) | 15 (21)
Epilepsy (Nervous system disorders) | 7 (8)
Status epilepticus (Nervous system disorders) | 5 (5)
Grand mal convulsion (Nervous system disorders) | 3 (3)
Headache (Nervous system disorders) | 2 (2)
Hydrocephalus (Nervous system disorders) | 2 (2)
Coordination abnormal (Nervous system disorders) | 2 (2)
Subarachnoid haemorrhage (Nervous system disorders) | 2 (2)
Monoparesis (Nervous system disorders) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1)
Cerebral haematoma (Nervous system disorders) | 1 (1)
Paresis (Nervous system disorders) | 1 (1)
Sciatica (Nervous system disorders) | 1 (1)
Visual field defect (Nervous system disorders) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 1 (1)
Complex partial seizures (Nervous system disorders) | 1 (1)
Encephalitis (Nervous system disorders) | 1 (1)
Aura (Nervous system disorders) | 1 (1)
Hemiparesis (Nervous system disorders) | 1 (1)
Intracranial pressure increased (Nervous system disorders) | 1 (1)
Simple partial seizures (Nervous system disorders) | 1 (1)
Depression (Psychiatric disorders) | 2 (2)
Epileptic psychosis (Psychiatric disorders) | 2 (3)
Aggression (Psychiatric disorders) | 1 (1)
Suicide attempt (Psychiatric disorders) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (1)
Pathological gambling (Psychiatric disorders) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1)
Calculus ureteric (Renal and urinary disorders) | 1 (1)
Metrorrhagia (Reproductive system and breast disorders) | 2 (2)
Ovarian cyst (Reproductive system and breast disorders) | 2 (2)
Bartholin's cyst (Reproductive system and breast disorders) | 1 (1)
Uterine polyp (Reproductive system and breast disorders) | 1 (1)
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bronchial disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Breast prosthesis user (Social circumstances) | 1 (1)
Shoulder operation (Surgical and medical procedures) | 1 (1)
Knee meniscectomy (Surgical and medical procedures) | 1 (1)
Hospitalisation (Surgical and medical procedures) | 1 (1)
Therapeutic procedure (Surgical and medical procedures) | 1 (1)
Ischaemia (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lacosamide (N=376)
Vertigo (Ear and labyrinth disorders) | 31 (35)
Diplopia (Eye disorders) | 51 (63)
Vomiting (Gastrointestinal disorders) | 25 (33)
Fatigue (General disorders) | 22 (25)
Nasopharyngitis (Infections and infestations) | 52 (77)
Contusion (Injury, poisoning and procedural complications) | 20 (29)
Back pain (Musculoskeletal and connective tissue disorders) | 28 (38)
Dizziness (Nervous system disorders) | 91 (157)
Headache (Nervous system disorders) | 54 (97)
Somnolence (Nervous system disorders) | 27 (34)
Tremor (Nervous system disorders) | 23 (31)
Balance disorder (Nervous system disorders) | 19 (25)
Convulsion (Nervous system disorders) | 19 (23)
Depression (Psychiatric disorders) | 19 (20)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
UCB has > 60 but <= 180 days to review results communications prior to public release and may delete information that is confidential and compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that the results shall be published regardless of outcome.